CLINICAL TRIAL: NCT00262015
Title: A Phase IV, Single Center, Open-Label, Controlled, Randomized Study to Evaluate the Memory Response of Children Previously Vaccinated With Chiron Meningococcal C Conjugate Vaccine, Menjugate® and Describe the Kinetic of the Antibody Response and Maturation on Days 2-7 and 28 After Challenge With Pasteur Merieux Meningococcal A/C Polysaccharide Vaccine or Menjugate®
Brief Title: Kinetic of Immune Memory Response After Re-Vaccination With Meningococcal Vaccine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chiron Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: M14P2
Record Dates: First submitted 2005-12-02; First posted 2005-12-06 (Estimated); Last update posted 2005-12-06 (Estimated); Status verified 2005-12

CONDITIONS: Meningococcal Disease; Meningococcal Meningitis
MeSH Terms: conditions — Meningococcal Infections; Meningitis, Meningococcal | interventions — serogroup C meningococcal conjugate vaccine

INTERVENTIONS:
Biological: · Meningococcal C conjugate vaccine; Meningococcal A/C Polysaccharide vaccine (partial dose)

SUMMARY:
The purpose of this study is to determine when a memory immune response after re-vaccination with Meningococcal C conjugate vaccine (Menjugate) or challenge with Meningococcal A/C polysaccharide vaccine can be observed, after initial vaccination with Meningococcal C conjugate vaccine during the UK immunization campaign

ELIGIBILITY:
Inclusion Criteria:

* Healthy adolescents between and including 13-15 years of age, who provide written informed consent and who received one immunization with Chiron Meningococcal C Conjugate vaccine (Menjugate) during the UK immunization campaign and for which documentation can be provided.

Exclusion Criteria:

* Subjects with a previous or suspected disease caused by N. meningitidis; or previous immunization with a meningococcal vaccine or vaccine containing meningococcal antigen(s); Any serious acute, chronic or progressive disease

Ages: 13 Years to 15 Years | Sex: All
Age Groups: Child
Enrollment: 264
Dates: Start 2003-09

PRIMARY OUTCOMES:
To measure immunological memory response to N. meningitidis serogroup C after those who received a partial dose of Meningococcal A/C Polysaccharide vaccine and in subjects who received a dose of Chiron Meningococcal C conjugate vaccine.

SECONDARY OUTCOMES:
To assess the immunological response to N. meningitidis serogroup C in those challenged with meningococcal A/C polysaccharide vaccine and in those who received a dose of Chiron Meningococcal C conjugate vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J. Pollard, MBBS, FRCPCH, PhD, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford, The Oxford Vaccine Group, Oxford, United Kingdom